CLINICAL TRIAL: NCT03250962
Title: Anti-PD-1 Antibody SHR-1210 Alone or in Combination With Decitabine in Relapsed or Refractory Hodgkin Lymphoma:an Open-label Phase II Trial
Brief Title: SHR-1210 Alone or in Combination With Decitabine in Relapsed or Refractory Hodgkin Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Principal Investigator, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-023
Record Dates: First submitted 2017-08-10; First posted 2017-08-16 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Hodgkin Lymphoma
Keywords: Relapsed/Refractory; Hodgkin Lymphoma；Decitabine; SHR-1210
MeSH Terms: conditions — Hodgkin Disease; Recurrence | interventions — camrelizumab; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1210-plus-Decitabine (Experimental): Decitabine 10 mg/day, days 1-5; SHR-1210 200 mg, day 8, every 3 weeks.
  Interventions: Drug: SHR-1210; Drug: Decitabine
- SHR-1210 (Experimental): SHR-1210 200 mg, day 1, every 3 weeks.
  Interventions: Drug: SHR-1210

INTERVENTIONS:
Drug: SHR-1210 — SHR-1210 is a humanized anti-PD-1 monoclonal antibody.
Drug: Decitabine — Decitabine is an investigational (experimental) drug that works by depleting DNA methyltransferase 1 (DNMT1), which can increase tumor antigens and HLA expression, enhances antigen processing, promotes T cell infiltration, and boosts effector T cell function.
  Arms: SHR-1210-plus-Decitabine

SUMMARY:
This is a two-stage, Phase II clinical trial for patients with relapsed or refractory Hodgkin Lymphoma. The purpose of stage I is to evaluate whether treatment with the study drug decitabine in combination with SHR-1210 is safe and more effective than treatment with SHR-1210 alone; and reverse the resistance of anti-PD-1 antibody in patients with HL who had previously treated with anti-PD-1 monotherapy. If it is deemed that the combination therapy is more efficacious than SHR-1210 monotherapy (The CR rate of the combination group is at least 30% higher compared to monotherapy group with a minimal follow-up of 6 months in predicting 60 subjects naïve to anti-PD-1 antibody who are randomly assigned (2:1) to the above two groups), the stage II study will be revised to a multicohort, decitabine-plus-SHR1210 single-arm clinical trial. The primary objective of stage II study is to evaluate the long-term response duration with decitabine-plus-SHR-1210 in relapsed or refractory Hodgkin Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* 1 Subjects must have histological confirmation of relapsed or refractory Hodgkin lymphoma (HL).

  2 12 to 75 years of age. 3 ECOG performance of less than 2. 4 Life expectancy of at least 3 months. 5 Subjects with lymphoma must have at least one measureable lesion >1 cm as defined by lymphoma response criteria.

  6 Subjects must have received at least four prior chemotherapy regimen, and must be off therapy for at least 4 weeks prior to Day 1. Subjects with autologous hematopoietic stem-cell transplantation are eligible which must be more than 3 months.Subjects with Anti-PD-1 antibody are eligible which must be resistance.

  7 Subjects must have adequate marrow, live, renal and heart functions.

Exclusion Criteria:

* 1 Subjects with any autoimmune disease or history of syndrome that requires corticosteroids or immunosuppressive medications.

  2 Serious uncontrolled medical disorders or active infections, pulmonary infection especially.

  3 Active alimentary tract hemorrhage or history of alimentary tract hemorrhage in 1 month .

  4 Prior organ allograft. 5 Women who are pregnant or breastfeeding. 6 Women with a positive pregnancy test on enrollment or prior to investigational product administration.

  7 Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2017-09-11 (Actual); Primary Completion 2022-07-21 (Estimated); Study Completion 2025-03-21 (Estimated)

PRIMARY OUTCOMES:
stage I: Number of Subjects with treatment-related adverse events (AEs) | 2 years
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v4.03.
stage I: CRR assess by investigators per the 2014 Lugano classification | 3 years
  rate of subjects achieved complete response in all evaluable subjects
stage II: duration of CR | 5 years
  Time measured from the day of first documented CR to the date of first documented progression, or death from any cause.

SECONDARY OUTCOMES:
stage II: duration of response | 5 years
  Time measured from the day of first documented PR or CR to the date of first documented progression, or death from any cause.
stage II: Progression free survival | 5 years
  Time measured from the day of treatment to the date of first documented progression, or death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Biotherapeutic Department of Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Study Protocol

REFERENCES:
- [Derived] Liu Y, Wang C, Li X, Dong L, Yang Q, Chen M, Shi F, Brock M, Liu M, Mei Q, Liu J, Nie J, Han W. Improved clinical outcome in a randomized phase II study of anti-PD-1 camrelizumab plus decitabine in relapsed/refractory Hodgkin lymphoma. J Immunother Cancer. 2021 Apr;9(4):e002347. doi: 10.1136/jitc-2021-002347. PMID 33820822
- [Derived] Wang C, Liu Y, Dong L, Li X, Yang Q, Brock MV, Mei Q, Liu J, Chen M, Shi F, Liu M, Nie J, Han W. Efficacy of Decitabine plus Anti-PD-1 Camrelizumab in Patients with Hodgkin Lymphoma Who Progressed or Relapsed after PD-1 Blockade Monotherapy. Clin Cancer Res. 2021 May 15;27(10):2782-2791. doi: 10.1158/1078-0432.CCR-21-0133. Epub 2021 Mar 5. PMID 33674274
- [Derived] Nie J, Wang C, Liu Y, Yang Q, Mei Q, Dong L, Li X, Liu J, Ku W, Zhang Y, Chen M, An X, Shi L, Brock MV, Bai J, Han W. Addition of Low-Dose Decitabine to Anti-PD-1 Antibody Camrelizumab in Relapsed/Refractory Classical Hodgkin Lymphoma. J Clin Oncol. 2019 Jun 10;37(17):1479-1489. doi: 10.1200/JCO.18.02151. Epub 2019 Apr 30. PMID 31039052